CLINICAL TRIAL: NCT06654531
Title: Comparative Study Between the Effect of Intravenous or Intrathecal Dexmedetomidine on Bupivacaine Spinal Block
Brief Title: Effect of Intravenous or Intrathecal Dexmedetomidine on Bupivacaine Spinal Block in Lower Abdominal Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, ahmed abed mansour, Dr, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 66
Record Dates: First submitted 2023-06-13; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2023-06

CONDITIONS: Spinal Anesthetics Causing Adverse Effects in Therapeutic Use
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: All patients will be assigned randomly into two groups :group 1 (the I.V group ) Patients in the I.V group (n = 25) received intrathecal hyperbaric bupivacaine 15 mg together with NSS 0.5 ml, followed by an I.V bolus dose of dexmedetomidine 0.5 μg/kg over 10 min and then an I.V infusion of a maintenance dose of 0.5 μg/kg/h (200 μg dexmedetomidine in 2 ml added to 48 ml NSS yielded dexmedetomidine 4 μg /ml) for the entire period of surgery.
  intrathecal group (n = 25) patients received intrathecal 15 mg hyperbaric bupivacaine together with 5 μg Dexmedetomidine 100 μg/ml diluted with normal saline solution (NSS) to 10 μg/ml), followed by an NSS I.V bolus and an I.V infusion of maintenance volume equivalent to that of the I.V group throughout the entire period of the surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- group 1 (I.V group ) (Active Comparator): Patients in the I.V group (n = 25) received intrathecal hyperbaric bupivacaine 15 mg together with NSS 0.5 ml, followed by an I.V bolus dose of dexmedetomidine 0.5 μg/kg over 10 min and then an I.V infusion of a maintenance dose of 0.5 μg/kg/h (200 μg dexmedetomidine in 2 ml added to 48 ml NSS yielded dexmedetomidine 4 μg /ml) for the entire period of surgery.
  Interventions: Drug: Dexmedetomidine
- group 2 (intrathecal group) (Active Comparator): 25 patients received intrathecal 15 mg hyperbaric bupivacaine (Marcaine 0.5%; Astra Zeneca, UK) together with 5 μg Dexmedetomidine (Precedex; Abbott; Chicago, IL, USA, 100 μg/ml diluted with normal saline solution (NSS) to 10 μg/ml), followed by an NSS I.V bolus and an I.V infusion of maintenance volume equivalent to that of the I.V group throughout the entire period of the surgery.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Under a sterile technique, spinal anesthesia will be carried out using a 22-G Quincke spinal needle after skin infiltration with 2% lidocaine 3 ml a t the L3-L4 level, a midline approach in the sitting position, and then in the supine position.
  Th e time of spinal injection will be considered time zero (T0). The I.V drug regimen will be started according to the group to which patients will be assigned.patients will receive intrathecal 15 mg hyperbaric bupivacaine together with 5 μg Dexmedetomidine in group 2

SUMMARY:
This study is a comparative study will be carried out after approval by the Local Ethical Committee in Al-Azhar University hospital (Assiut) and after obtaining patients' written informed consent.

50 ASA physical status I-II aged 20-60 years of both sexes scheduled for lower abdominal surgery with an expected duration of 90-120 min under spinal anesthesia will be enrolled in this study

Primary outcome :

- The onset and duration of sensory and motor blockade ,Postoperative analgesic efficacy .

Secondary outcomes :

- to assess the effect on hemodynamics and postoperative analgesic requirement All patients will be assigned randomly into two groups :group 1 (the I.V group ) Patients in the I.V group (n = 25) received intrathecal hyperbaric bupivacaine 15 mg together with NSS 0.5 ml, followed by an I.V bolus dose of dexmedetomidine 0.5 μg/kg over 10 min and then an I.V infusion of a maintenance dose of 0.5 μg/kg/h (200 μg dexmedetomidine in 2 ml added to 48 ml NSS yielded dexmedetomidine 4 μg /ml) for the entire period of surgery. intrathecal group (n = 25) patients received intrathecal 15 mg hyperbaric bupivacaine (Marcaine 0.5%; Astra Zeneca, UK) together with 5 μg Dexmedetomidine (Precedex; Abbott; Chicago, IL, USA, 100 μg/ml diluted with normal saline solution (NSS) to 10 μg/ml), followed by an NSS I.V bolus and an I.V infusion of maintenance volume equivalent to that of the I.V group throughout the entire period of the surgery.

DETAILED DESCRIPTION:
Neuraxial anesthesia and analgesia provide a solid analgesic effect by inhibiting nociceptive transmission from peripheral to the central neuronal system . However, their analgesic advantages might be limited by the short life of current local anesthetics (LAs). Therefore, adjunct analgesic strategy is an alternative to prolonging the analgesic duration and decreases the potential risk of side effects by reducing the dose of LA.

This study is a comparative study will be carried out after approval by the Local Ethical Committee in Al-Azhar University hospital (Assiut) and after obtaining patients' written informed consent. inclusion criteria will be: 50 ASA physical status I-II aged 20-60 years of both sexes scheduled for lower abdominal surgery with an expected duration of 90-120 min under spinal anesthesia will be enrolled in this study. Exclusion criteria

* Patient refusal.
* history of cardiac, hepatic, neurological, or renal disease.
* BMI ≥30kg/ m2 (Morbid obesity).
* Patients with diabetes mellitus.
* history of allergy to study drugs, any contraindication for regional anesthesia
* Coagulopathy.
* failed or unsatisfactory spinal block. Study tools All patients will be assigned randomly into two groups :group 1 (the I.V group ) Patients in the I.V group (n = 25) received intrathecal hyperbaric bupivacaine 15 mg together with NSS 0.5 ml, followed by an I.V bolus dose of dexmedetomidine 0.5 μg/kg over 10 min and then an I.V infusion of a maintenance dose of 0.5 μg/kg/h (200 μg dexmedetomidine in 2 ml added to 48 ml NSS yielded dexmedetomidine 4 μg /ml) for the entire period of surgery.

intrathecal group (n = 25) patients received intrathecal 15 mg hyperbaric bupivacaine together with 5 μg Dexmedetomidine100 μg/ml diluted with normal saline solution (NSS) to 10 μg/ml), followed by an NSS I.V bolus and an I.V infusion of maintenance volume equivalent to that of the I.V group throughout the entire period of the surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II
* lower abdominal surgery
* Aged 20-60 years of both sexes

Exclusion Criteria:

* Patient refusal.
* history of cardiac, hepatic, neurological, or renal disease.
* BMI ≥30kg/ m2 (Morbid obesity).
* Patients with diabetes mellitus.
* history of allergy to study drugs, any contraindication for regional anesthesia
* Coagulopathy.
* failed or unsatisfactory spinal block.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
Postoperative analgesic efficacy | 15 minutes intervals for 12 hours postoperatively
  duration of sensory blockade of spinal anaesthesia
Postoperative analgesic efficacy | 20 minutes intervals for 12 hours postoperatively
  duration of motor blockade of spinal anesthesia

SECONDARY OUTCOMES:
Haemodynamics | 1 hours intervals from start of operation until 12 hours postoperatively
  heart rate
Assessment of pain | every 1 hour intervals until 12 hours postoperatively
  NRS 0-10 (0 = no pain, 10 = the worst pain imaginable)
Assessment of sedation | every 30 minutes intervals for 12 hours postoperatively
  Ramsay sedation scale
hemodynamics | 1 hours intervals from start of operation until 12 hours postoperatively
  Mean blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: ezzat m ali el soudy, professor, Study Chair — professor of anaesthesia and icu
Locations (1):
- Azhar University, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
analytical data will be available